CLINICAL TRIAL: NCT02238028
Title: Short-term Cardiovascular Benefits of Wearing Particulate-filtering Respirators: a Randomized Controlled Crossover Trial Among Healthy Young Adults
Brief Title: Short-term Cardiovascular Benefits of Wearing Particulate-filtering Respirators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haidong Kan, Professor, Ph.D., Fudan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: KZGY 001
Record Dates: First submitted 2014-09-07; First posted 2014-09-12 (Estimated); Results first posted 2016-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-04

CONDITIONS: Autonomic Nervous System Imbalance; Blood Pressure; Inflammation; Vasoconstriction; Blood Coagulation Disorders
Keywords: Heart rate variability; Blood pressure; Circulating biomarkers; Respirator; Fine particulate matter
MeSH Terms: conditions — Inflammation; Blood Coagulation Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wear respirator (Experimental): The recruited healthy subjects were randomly allocated into two groups.In each intervention, one group wore the high-efficiency respirator as much as possible for continuous 48hr and the other group behaved as usual. After a three-week interval, the two groups exchanged their roles in wearing the respirator or not. The same protocol on the measurements of health indicators and ambient air pollution was applied in the 1st intervention and 2nd intervention period.
  Interventions: Behavioral: Wear respirator
- Not wear respirator (No Intervention): The recruited healthy subjects were randomly allocated into two groups.In each intervention, one group wore the high-efficiency respirator as much as possible for continuous 48hr and the other group behaved as usual. After a three-week interval, the two groups exchanged their roles in wearing the respirator or not. The same protocol on the measurements of health indicators and ambient air pollution was applied in the 1st intervention and 2nd intervention period.

INTERVENTIONS:
Behavioral: Wear respirator — Healthy adult subjects wore the particulate filtering respirators for continuous 48 hours as much as possible both indoor and outdoor.
  Other Names: particulate filtering respirator
  Arms: Wear respirator

SUMMARY:
An intervention study to assess the short-term cardiovascular effects of reducing personal air pollution exposure by wearing particulate filtering respirators.

DETAILED DESCRIPTION:
A group of healthy adult college students fulfilling the recruitment criteria were randomly divided into two sub-groups. One sub-group weared the particulate filtering respirators for 2 continuous days during which the respirator was required to wear as much as possible both indoor and outdoor. The other group acted as normal at the same time. The measurements on health effects including heart rate varibility, blood pressure, circulating biomarkers as well as the ambient air pollution were performed in both groups during the intervention period. After a 3-week rest period,the two groups interchanged their roles of wearing the respirator or not. The same measurements of both health effects indicators and ambient air pollution were repeated.

ELIGIBILITY:
Inclusion Criteria:

* Equal to or older than 18 years old,
* No history of smoking and alcohol addiction.
* No chronic diseases,such as hypertension,diabetes,chronic obstructive pulmonary disease or other respiratory/cardiovascular diseases reported by volunteers.
* No respiratory or allergic diseases, like asthma, rhinitis,or other allergic diseases.

Exclusion Criteria:

* Current smokers
* Chronic drug use due on cardiovascular or respiratory diseases

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kan Haidong, PhD, Study Director — School of Public Health，Fudan University
Locations (1):
- Department of Environmental Health, School of Public Health, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Shah AS, Langrish JP, Nair H, McAllister DA, Hunter AL, Donaldson K, Newby DE, Mills NL. Global association of air pollution and heart failure: a systematic review and meta-analysis. Lancet. 2013 Sep 21;382(9897):1039-48. doi: 10.1016/S0140-6736(13)60898-3. Epub 2013 Jul 10. PMID 23849322
- [Background] Chen R, Zhao A, Chen H, Zhao Z, Cai J, Wang C, Yang C, Li H, Xu X, Ha S, Li T, Kan H. Cardiopulmonary benefits of reducing indoor particles of outdoor origin: a randomized, double-blind crossover trial of air purifiers. J Am Coll Cardiol. 2015 Jun 2;65(21):2279-87. doi: 10.1016/j.jacc.2015.03.553. PMID 26022815

RESULTS

PARTICIPANT FLOW:
Groups:
- Wearing Respirator First,Then Not Wearing Respirator: The recruited healthy subjects were randomly allocated into two groups. In the first intervention period, this group wore respirator for 2 continuous days. After a 3-week washout period, the 2nd intervention period started and they changed to not wearing the respirator but participated all the measurements of health indicators and ambient air pollution for 2 continuous days. The same protocol on the measurements of health indicators and ambient air pollution was applied in the 1st intervention and 2nd intervention period.
  Wear respirator: Healthy adult subjects wore the particulate filtering respirators for continuous 48 hours as much as possible both indoor and outdoor.
- Not Wearing Respirator First,Then Wearing Respirator: The recruited healthy subjects were randomly allocated into two groups. In the first intervention period, this group did not wear respirator but participated all the measurements on health indicator and ambient air pollution for 2 continuous days. After a 3-week washout period, the 2nd intervention period started and they changed to wear the respirator for 2 continuous days. The same protocol on the measurements of health indicators and ambient air pollution was applied in the 1st intervention and 2nd intervention period.
Period: Overall Study
Arm/Group | Wearing Respirator First,Then Not Wearing Respirator | Not Wearing Respirator First,Then Wearing Respirator
Started | 14 | 14
Completed | 12 | 12
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: The recruited healthy subjects were randomly allocated into two groups. In the first intervention period, this group wore respirator for 2 continuous days including a 2-hour walking along the streets on the 2nd day along a fixed route. After a 2-week rest period, the 2nd intervention period started and they changed to not wearing the respirator but participated all the measurements of health indicators and ambient air pollution for 2 continuous days including the 2-hour walking along the streets on the 2nd day along the same fixed route. The same protocol on the measurements of health indicators and ambient air pollution was applied in the 1st intervention and 2nd intervention period.
  Wear respirator: Healthy adult subjects wore the particulate filtering respirators for continuous 48 hours as much as possible both indoor and outdoor.
Arm/Group | All Study Participants
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13
Region of Enrollment [Number; unit: participants]
  China | 24
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22 (4)
systolic pressure [Mean (Standard Deviation); unit: mmHg] | 108 (8)
diastolic pressure [Mean (Standard Deviation); unit: mmHg] | 70 (5)

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate Variability-LF Power,HF Power,VLF Power
Description: HRV is a quantitative health marker reflecting how the autonomic nervous system modulates the sinoatrial node in the heart and HRV has therefore been widely used to estimate cardiac autonomic function and control. Subjects were attached with Holter monitor on the 2nd day in each of the 48-hr intervention period.A total of 8 parameters of HRV were analyzed including 4 time-domain indices and 4 frequency-domain indices. Frequency domain methods assign bands of frequency and then count the number of NN intervals that match each band. The bands are typically high frequency (HF) from 0.15 to 0.4 Hz, low frequency (LF) from 0.04 to 0.15 Hz, and the very low frequency (VLF) from 0.0033 to 0.04 Hz. Parasympathetic activity is a major contributor to the HF component. More problematic is the interpretation of the LF component, which was considered by some as a marker of sympathetic modulation but is now known to include both sympathetic and vagal influences.
Time Frame: up to 24 hours
Measure: Geometric Mean (Standard Deviation); unit: ms^2
Groups:
- Wear Respirator: The subjects were randomized into 2 groups. In each intervention, one group wore the high-efficiency respirator as much as possible for continuous 48hr and the other group behaved as usual. After a three-week interval, the two groups exchanged their roles in wearing the respirator or not. The same protocol on the measurements of health indicators and ambient air pollution was applied in the 1st intervention and 2nd intervention period.
  Wear respirator: Healthy adult subjects wore the particulate filtering respirators for continuous 48 hours as much as possible both indoor and outdoor.
- Not Wear Respirator: The subjects were randomized into 2 groups. In each intervention, one group wore the high-efficiency respirator as much as possible for continuous 48hr and the other group behaved as usual. After a three-week interval, the two groups exchanged their roles in wearing the respirator or not. The same protocol on the measurements of health indicators and ambient air pollution was applied in the 1st intervention and 2nd intervention period.
Arm/Group | Wear Respirator | Not Wear Respirator
Number analyzed (Participants) | 24 | 24
ms^2
  low frequency(LF) power | 899.4 (601.3) | 838.5 (562.4)
  high frequency(HF) power | 519.7 (371.0) | 416.6 (296.6)
  very low frequency(VLF) power | 1684.6 (875.7) | 1623.1 (1006.5)
Statistical Analysis 1: Comparison: Wear Respirator vs Not Wear Respirator; Paired Student's t tests were used in the absence and presence of wearing respirators. HRV was log-transformed before regression analyses. Linear mixed-effect models were applied to investigate the effects of wearing respirators. Age, sex, body mass index, PM2.5 concentration, 48-h mean temperature and 48-h mean humidity were introduced into the model as fixed-effect terms. At last, we incorporated random-effect intercepts for subjects to account for correlations between repeated measurements; Test type: Superiority or Other; p < 0.05, Paired t-test,2 sided

2. Primary Outcome: Blood Pressure
Description: The blood pressure were measured by automatic blood pressure monitor during the intervention study.
Time Frame: up to 24 hours
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Wear Respirator | Not Wear Respirator
Number analyzed (Participants) | 24 | 24
mmHg
  systolic blood pressure | 107.3 (8.0) | 109.0 (7.4)
  diastolic blood pressure | 70.0 (5.0) | 70.8 (4.8)
Statistical Analysis 1: Comparison: Wear Respirator vs Not Wear Respirator; Test type: Superiority or Other; p < 0.05, Paired t-test,2 sided

3. Primary Outcome: Heart Rate Variability-SDNN,SDANN, rMSSD
Description: HRV is a quantitative health marker reflecting how the autonomic nervous system modulates the sinoatrial node in the heart and HRV has therefore been widely used to estimate cardiac autonomic function and control.A total of 8 parameters of HRV were analyzed including 4 time-domain indices and 4 frequency-domain indices. Subjects were attached with Holter monitor on the 2nd day in each of the 48-hr intervention period. Heart rate and heart automatic function indices including the standard deviation of the normal-to-normal interval(SDNN),the standard deviation of the average NN intervals calculated over short periods(SDANN), the root mean square of the successive differences(rMSSD) were automatically recorded during the intervention.
Time Frame: Up to 24 hours
Measure: Geometric Mean (Standard Deviation); unit: ms
Groups:
- All Study Participants: The recruited healthy subjects were randomly allocated into two groups. In the first intervention period, this group wore respirator for 2 continuous days. After a 3-week washout period, the 2nd intervention period started and they changed to not wearing the respirator but participated all the measurements of health indicators and ambient air pollution for 2 continuous days. The same protocol on the measurements of health indicators and ambient air pollution was applied in the 1st intervention and 2nd intervention period.
  Wear respirator: Healthy adult subjects wore the particulate filtering respirators for continuous 48 hours as much as possible both indoor and outdoor.
Arm/Group | All Study Participants
Number analyzed (Participants) | 24
ms
  SDNN | 177.5 (29.9)
  SDANN | 160.7 (28.9)
  rMSSD | 49.0 (13.3)

4. Primary Outcome: Heart Rate Variability-LF/HF
Description: HRV is a quantitative health marker reflecting how the autonomic nervous system modulates the sinoatrial node in the heart and HRV has therefore been widely used to estimate cardiac autonomic function and control. Subjects were attached with Holter monitor on the 2nd day in each of the 48-hr intervention period.A total of 8 parameters of HRV were analyzed including 4 time-domain indices and 4 frequency-domain indices. Frequency domain methods assign bands of frequency and then count the number of NN intervals that match each band. The bands are typically high frequency (HF) from 0.15 to 0.4 Hz, low frequency (LF) from 0.04 to 0.15 Hz. Parasympathetic activity is a major contributor to the HF component. More problematic is the interpretation of the LF component, which was considered by some as a marker of sympathetic modulation but is now known to include both sympathetic and vagal influences.
Time Frame: Up to 24 hours
Measure: Geometric Mean (Standard Deviation); unit: ratio
Groups:
- Wear Respirator: The recruited healthy subjects were randomly allocated into two groups. In the first intervention period, this group wore respirator for 2 continuous days. After a 3-week washout period, the 2nd intervention period started and they changed to not wearing the respirator but participated all the measurements of health indicators and ambient air pollution for 2 continuous days. The same protocol on the measurements of health indicators and ambient air pollution was applied in the 1st intervention and 2nd intervention period.
  Wear respirator: Healthy adult subjects wore the particulate filtering respirators for continuous 48 hours as much as possible both indoor and outdoor.
- Not Wear Respirator: The recruited healthy subjects were randomly allocated into two groups. In the first intervention period, this group did not wear respirator but participated all the measurements on health indicator and ambient air pollution for 2 continuous days. After a 3-week washout period, the 2nd intervention period started and they changed to wear the respirator for 2 continuous days. The same protocol on the measurements of health indicators and ambient air pollution was applied in the 1st intervention and 2nd intervention period.
Arm/Group | Wear Respirator | Not Wear Respirator
Number analyzed (Participants) | 24 | 24
ratio | 1.4 (0.3) | 1.5 (0.3)

5. Primary Outcome: Heart Rate Variability-pNN50
Description: HRV is a quantitative health marker reflecting how the autonomic nervous system modulates the sinoatrial node in the heart and HRV has therefore been widely used to estimate cardiac autonomic function and control.A total of 8 parameters of HRV were analyzed including 4 time-domain indices and 4 frequency-domain indices. Subjects were attached with Holter monitor on the 2nd day in each of the 48-hr intervention period. Heart rate and heart automatic function indices including the proportion of successive normal NN intervals differing by more than 50 ms in the total number of NNs（pNN50） were automatically recorded during the intervention.
Time Frame: Up to 24 hours
Measure: Geometric Mean (Standard Deviation); unit: percentage of ms
Arm/Group | Wear Respirator | Not Wear Respirator
Number analyzed (Participants) | 24 | 24
percentage of ms | 24.0 (9.9) | 20.5 (10.5)

6. Primary Outcome: Circulating Biomarkers--Fibrinogen，vWF
Description: At the end of each intervention, participants were asked to rest in a quiet room for half an hour. Peripheral venous blood samples were collected and centrifuged immediately. The serum were collected and stored at -80℃ within 30 minutes to minimize the in-vitro changes in biomarker proteins. Fibrinogen and von Willebrand factor(vWF) were measured by using the Millipore MILLIPLEX MAP human cytokine/chemokine kit (Millipore Corp., Billerica, Massachusetts)
Time Frame: Up to 24 hours
Measure: Geometric Mean (Standard Deviation); unit: µg/ml
Arm/Group | Wear Respirator | Not Wear Respirator
Number analyzed (Participants) | 24 | 24
µg/ml
  Fibrinogen | 2.5 (1.3) | 2.5 (1.3)
  vWF | 24.5 (1.3) | 27.1 (1.3)

7. Primary Outcome: Circulating Biomarkers--P- Selectin,VCAM-1
Description: At the end of each intervention, participants were asked to rest in a quiet room for half an hour. Peripheral venous blood samples were collected and centrifuged immediately. The serum were collected and stored at -80℃ within 30 minutes to minimize the in-vitro changes in biomarker proteins. P- selectin,VCAM-1(vascular cell adhesion molecule-1) were measured by using the Millipore MILLIPLEX MAP human cytokine/chemokine kit (Millipore Corp., Billerica, Massachusetts)
Time Frame: Up to 24 hours
Measure: Geometric Mean (Standard Deviation); unit: ng/ml
Arm/Group | Wear Respirator | Not Wear Respirator
Number analyzed (Participants) | 24 | 24
ng/ml
  P-selectin | 164.0 (2.0) | 200.3 (1.5)
  VCAM-1 | 1480.3 (1.5) | 1808.0 (1.6)

8. Primary Outcome: Circulating Biomarkers--ET-1
Description: At the end of each intervention, participants were asked to rest in a quiet room for half an hour. Peripheral venous blood samples were collected and centrifuged immediately. The serum were collected and stored at -80℃ within 30 minutes to minimize the in-vitro changes in biomarker proteins. Endothelin-1(ET-1) was using enzyme-linked immunosorbent assays.
Time Frame: Up to 24 hours
Measure: Geometric Mean (Standard Deviation); unit: pg/ml
Arm/Group | Wear Respirator | Not Wear Respirator
Number analyzed (Participants) | 24 | 24
pg/ml | 109.9 (1.6) | 121.5 (1.6)

ADVERSE EVENTS:
Time Frame: At the end of each 2-day period
Arm/Group | Wear Respirator | Not Wear Respirator
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes